CLINICAL TRIAL: NCT03110549
Title: A Phase 1, Randomized, Double-Blinded, Placebo-Controlled, Sequential Single Dose Escalation Study of the Safety, Tolerability and Pharmacokinetics of Subcutaneously and Intramuscularly Administered TMB-607 in HIV-Negative Volunteers
Brief Title: Study of the Safety, Tolerability and Pharmacokinetics of TMB-607 in HIV-Negative Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug development suspended by current holder of IND
Sponsor: TaiMed Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: TMB 607 101
Record Dates: First submitted 2017-03-31; First posted 2017-04-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Five qualifying participants will be enrolled into each of seven dosage Arms - three escalating subcutaneous dosages (Cohort 1), and four escalating intramuscular dosages (Cohort 2). Enrolling participants will be randomized to receive active TMB-607 or placebo. Beginning with the lowest dosage group, a Data Safety Monitoring Board (DSMB) will review available data after four participants have completed two weeks of post-dose follow-up to determine whether escalation to the next dosage group may proceed
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Cohort 1 Arm A (Experimental): Subcutaneous 200 mg of TMB-607 on Day 0 or Placebo
  Interventions: Drug: TMB-607; Drug: Placebo
- Cohort 1 Arm B (Experimental): Subcutaneous 500 mg of TMB-607 on Day 0 or Placebo
  Interventions: Drug: TMB-607; Drug: Placebo
- Cohort 1 Arm C (Experimental): Subcutaneous 1000 mg of TMB-607 on Day 0 or Placebo
  Interventions: Drug: TMB-607; Drug: Placebo
- Cohort 2 Arm A (Experimental): Subcutaneous 100 mg of TMB-607 on Day 0 or Placebo
  Interventions: Drug: TMB-607; Drug: Placebo
- Cohort 2 Arm B (Experimental): Subcutaneous 400 mg of TMB-607 on Day 0 or Placebo
  Interventions: Drug: TMB-607; Drug: Placebo
- Cohort 2 Arm C (Experimental): Subcutaneous 800 mg of TMB-607 on Day 0 or Placebo
  Interventions: Drug: TMB-607; Drug: Placebo
- Cohort 2 Arm D (Experimental): Subcutaneous 1500 mg of TMB-607 on Day 0 or Placebo
  Interventions: Drug: TMB-607; Drug: Placebo

INTERVENTIONS:
Drug: TMB-607
Drug: Placebo

SUMMARY:
The study is a Phase 1, randomized, double-blinded, placebo-controlled, sequential single dose escalation safety, tolerability and pharmacokinetic study of subcutaneous and intramuscular TMB-607 administered to HIV-negative volunteers.

DETAILED DESCRIPTION:
This study uses a sequential dose-escalation design for single dose subcutaneous and intramuscular administrations in HIV-negative volunteers. The study investigates seven TMB-607 dose groups: Cohort 1: 200 mg subcutaneously (Arm A), 500 mg subcutaneously (Arm B) and 1,000 mg subcutaneously (Arm C); Cohort 2: 100 mg intramuscularly (Arm A), 400 mg intramuscularly (Arm B), 800 mg intramuscularly (Arm C) and 1,500 mg intramuscularly (Arm D). Five participants will be enrolled in each dose group, and will be randomly assigned in a 4:1 ratio to receive TMB-607 or placebo in a double-blinded fashion (four participants per group assigned to active TMB-607; one participant per group assigned to placebo). In each group, a single dose injection of TMB-607 or placebo will be administered at Day 0. The first three Day 0 injections administered in each dose group must be given at least 24 hours apart. Subjects will be enrolled sequentially so that a maximum of three subjects in each Cohort is dosed within any 24-hour period. All subjects will be monitored for 24 hours after study drug administration, with vital signs and ECGs checked hourly, and intensive pharmacokinetic samples collected during this period. Study drug will only be administered on Mondays to prevent weekend days from interfering with the daily assessments closest to the time of dosing. Participants will be followed for 10 weeks after receiving study drug.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following criteria to be included in the study:

  1. Male or female between 18-55 years of age on the day of screening
  2. HIV-negative volunteers, willing to undergo HIV testing and counseling, and receive HIV test results
  3. Normal 12-lead ECG at Screening and on Day 0, including normal sinus rate and rhythm, QTc interval ≤440msec, PR interval ≤200msec, and lack of any evidence of heart block, or left or right bundle branch block
  4. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study
  5. In the opinion of the principal investigator or designee, has understood the information provided; written informed consent needs to be given before any study-related procedures are performed
  6. Agrees to use a barrier form of contraception if engaging in sexual activity at any time throughout the study (males and females) - two reliable forms of barrier contraception diaphragm, Intra Uterine Device (IUD), spermicides or condoms) must be used if participants engage in sexual activity that could result in pregnancy; hormonal contraception (e.g., oral contraceptive pill, injectable or implantable contraceptive) must not be relied upon while in this study; all female participants must be willing to undergo urine pregnancy tests at time points indicated in the Schedule of Events and Procedures
  7. For females of reproductive potential, negative urine pregnancy test at screening and within 96 hours prior to randomization; female participants of reproductive potential are defined as women who have not been post-menopausal for at least 24 consecutive months (i.e., who have had menses within the preceding 24 months) or have not undergone surgical sterilization (e.g., hysterectomy, or bilateral oophorectomy, salpingectomy, or tubal ligation)

Exclusion Criteria:

* Participants having or meeting any of the following conditions or characteristics will be excluded from the study:

  1. Confirmed HIV-1 or HIV-2 infection
  2. Currently pregnant or breastfeeding
  3. Known allergy/sensitivity or any hypersensitivity to components of study drug or its formulation, or known allergy to sulfonamide drugs
  4. History, or family history of Short of Long QT syndrome, Wolff-Parkinson-White Syndrome, or congenital heart disease
  5. Family history of sudden cardiac death, or unexplained cardiac death in an otherwise healthy individual between the ages of 1 and 40 years
  6. History of syncope, palpitations, unexplained dizziness, hypokalemia, heart arrhythmias, or significant cardiac disease
  7. Major psychiatric illness including any history of schizophrenia or severe psychosis, bipolar disorder requiring therapy, suicide attempt in the previous 3 years
  8. Serious illness requiring systemic treatment and/or hospitalization within 21 days prior to randomization
  9. Receipt of immunomodulatory agents (e.g., interleukins, interferons, cyclosporine, systemic corticosteroids), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 180 days prior to study entry
  10. Any clinically significant acute or chronic medical condition requiring care of a physician (e.g., diabetes, coronary artery disease, rheumatologic illness, malignancy, substance abuse) that in the opinion of the investigator would preclude participation
  11. Any laboratory value of Grade 1 or higher according to the NCI Common Toxicity Criteria (Appendix A)
  12. Confirmed diagnosis of hepatitis B (surface antigen, HbsAg), or hepatitis C (HCV antibodies)
  13. Current confirmed STD infection
  14. In the opinion of the investigator, unlikely to comply with protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
TMB 607 plasma concentrations | 10 Weeks Post Injection
  Measurements of concentrations of TMB-607 in plasma will be used to determine the concentration-time profile of subcutaneous and intramuscular TMB-607 in all participants. TMB-607 plasma concentrations will be measured by a central lab using high-performance liquid chromatography - mass (HPLC-MS) method validated for the measurement of TMB-607 in human plasma.

SECONDARY OUTCOMES:
Adverse Events Related to Treatment | 10 Weeks Post Injection
  The frequency of adverse events will be tabulated by the Medical Dictionary for Regulatory Activities (MedDRA) term and system organ class. The maximum intensity and frequency of adverse events will be summarized by treatment group

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Jacobson, MD, Principal Investigator — Lewis Katz School of Medicine at Temple University
Locations (1):
- Lewis Katz School of Medicine at Temple University, Philadelphia, Pennsylvania, United States